CLINICAL TRIAL: NCT03964090
Title: A Study of Temozolomide, Etoposide, Doxil, Dexamethasone, Ibrutinib, and Rituximab (TEDDI-R) in Aggressive B-cell Lymphomas With Secondary Involvement of the Central Nervous System (CNS)
Brief Title: Temozolomide, Etoposide, Doxil, Dexamethasone, Ibrutinib, and Rituximab (TEDDI-R) in Aggressive B-cell Lymphomas With Secondary Involvement of the Central Nervous System (CNS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190103; 19-C-0103
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12-12

CONDITIONS: Central Nervous System Lymphoma; Secondary Central Nervous System Lymphoma
Keywords: Tyrosine Kinase Inhibitor; Lymphoma in Brain and CNS; ABC DLBCL; Diffuse Large B-Cell Lymphomas in CNS
MeSH Terms: interventions — ibrutinib; Cytarabine; isavuconazole; Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Temozolomide, etoposide, doxil, dexamethasone, and rituximab without ibrutinib (TEDD-R) or TEDD-R with ibrutinib (TEDDI-R), concurrent with cytarabine and isavuconazole, based upon response to 14-day ibrutinib window
  Interventions: Drug: TEDD-R; Drug: TEDDI-R; Drug: Ibrutinib; Drug: Cytarabine; Drug: Isavuconazole
- 2 (Experimental): Temozolomide, etoposide, doxil, dexamethasone, and rituximab without ibrutinib (TEDD-R) or TEDD-R with ibrutinib Days 1-10 (TEDDI-R), concurrent with cytarabine and isavuconazole, based upon response to 14-day ibrutinib window
  Interventions: Drug: TEDD-R; Drug: TEDDI-R; Drug: Ibrutinib; Drug: Cytarabine; Drug: Isavuconazole; Drug: Methotrexate

INTERVENTIONS:
Drug: TEDD-R — Temozolomide, etoposide, doxil, dexamthasone, and rituximab (TEDD-R) given every 21 days for cycles 1-4
Drug: TEDDI-R — Temozolomide, etoposide, doxil, dexamthasone, ibrutinib and rituximab (TEDDI-R) given every 21 days for cycles 1-4
Drug: Ibrutinib — For Arm 1:Ibrutinib given on days -14 to day -1 prior to cycle 1;then given every 21 days for cycles 1-4 For Arm 2: Ibrutinib given on days -14 to day -1 prior to cycle 1; then on days 1-10 for cycles 1-4
Drug: Cytarabine — Cytarabine on days 1 and day 5 of cycles 2-5 (all arms), as applicable
Drug: Isavuconazole — Isavuconazole to begin at least 3 days prior to ibrutinib and continue throughout chemotherapy unless ibrutinib discontinued permanently
Drug: Methotrexate — Methotrexate on days 1 and day 5 of cycles 2-5 (all arms), as applicable
  Arms: 2

SUMMARY:
Background:

Secondary central nervous system lymphoma (sCNSL) is cancer that has spread to the central nervous system. Most drugs used to treat it do not cross the blood-brain barrier. This makes it hard to treat. Researchers hope that a new combination of drugs may be able to help.

Objective:

To find a better way to treat sCNSL.

Eligibility:

People ages 18 and older with sCNSL

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood, urine, and heart tests
* Eye exam
* Tissue or tumor biopsy
* Collection of cerebrospinal fluid
* CT, PET, and MRI scans: Participants will like in a machine that takes pictures of the body.
* Bone marrow aspirations or biopsies: A needle will be inserted into the participant s hipbone. The needle will remove a small amount of marrow.

Participants will take the study drugs in 21-day cycles. They will take some drugs by mouth. They will take others through a catheter: A small tube will be inserted into a vein in the arm, neck, or chest. They may have drugs given through a catheter placed through the brain or injected into the spinal canal.

Participants will have regular visits during the study. These will include repeats of the screening test. They may also provide a saliva sample or have a cheek swab.

Participants will have up to 4 treatment cycles.

Participants will have a follow-up visit 30 days after their last treatment dose. Then they will have visits every 3-6 months for 3 years and then yearly....

DETAILED DESCRIPTION:
Background:

* Aggressive B-cell lymphomas with secondary involvement of the CNS (sCNSL) have a grave prognosis
* No standard of care exists for sCNSL; treatment approaches include combination chemotherapy regimens effective in primary CNS lymphoma (PCNSL)
* Ibrutinib is an inhibitor of Bruton s tyrosine kinase (BTK) and has demonstrated a high response rate in PCNSL and sCNSL but with short response duration
* We developed a novel regimen that combines ibrutinib with a chemoimmunotherapy platform maximized for CNS penetrance that includes temozolomide, etoposide, Doxil, dexamethasone, and rituximab (TEDDI-R) for aggressive B-cell lymphomas in the CNS
* A phase 1 study of TEDDI-R demonstrated durable remissions in refractory PCNSL
* We propose a small phase 2 to study the safety and efficacy of TEDDI-R in sCNSL

Objective:

-To estimate the progression-free survival (PFS) after TEDDI-R or TEDD-R in secondary CNS lymphoma (sCNSL)

Eligibility:

* Aggressive B-cell lymphomas with secondary involvement of the CNS (sCNSL)
* Relapsed/refractory from prior therapy or untreated with CNS involvement
* Age greater than or equal to 18 years
* No pregnant or nursing women
* Adequate organ function (defined in protocol)

Design:

* Phase II study of 58 evaluable participants with untreated and relapsed/refractory sCNSL (accrual ceiling will be set at 61 to allow for a few possible inevaluable participants)
* Participants will first be treated with a 14-day "window" of ibrutinib monotherapy in combination with isavuconazole to establish efficacy of ibrutinib. Participants who are known refractory to BTK inhibitors will skip the 14-day and proceed on to chemotherapy.
* Following the 14-day ibrutinib window, participants with at least a 20% reduction in bidimensional masses on imaging scans or those without measurable disease will receive ibrutinib with TEDD-R (TEDDI-R) chemotherapy for 4 cycles. Participants who are previously known to be refractory to BTK inhibitors and those who have less than a 20% reduction during the ibrutinib window will receive TEDD-R (without ibrutinib) for 4 cycles.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed secondary involvement of an aggressive B-cell lymphoma in the CNS (eye, CSF, and/or brain parenchyma).

NOTE: B-cell lymphomas that were previously indolent but now involve the CNS (i.e. transformed from previous follicular lymphoma or chronic lymphocytic leukemia and mantle cell lymphoma) are eligible.

* Participants must have disease that is relapsed or refractory after initial systemic treatment or participants without prior therapy for systemic DLBCL must have concomitant involvement of the eyes, CSF or brain parenchyma.
* Age greater than or equal to18 years. NOTE: Because no dosing or adverse event data are currently available on the use of ibrutinib and TEDDI-R in participants <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
* ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%) unless due to disease
* Participants must have adequate organ function as defined below, independent of growth factor or platelet transfusion support:

  * Absolute neutrophil count (ANC): greater than or equal to 750 cells/mcL (0.75 (SqrRoot) 10^9/L)
  * Platelets: greater than or equal to 50,000 cells/mcL (50 (SqrRoot) 10^9/L)
  * Hemoglobin: greater than or equal to 8 g/dL (transfusions permitted)
  * Serum total bilirubin: less than or equal to 1.5 X ULN unless Gilbert s syndrome or disease infiltration of the liver is present)
  * AST (SGOT) and ALT (SGPT): less than or equal to 3.0 (SqrRoot) institutional ULN (less than or equal to 5 x ULN for participants with liver involvement by lymphoma)
  * Serum creatinine: less than or equal to 1.5 mg/dL OR
  * Creatinine clearance: greater than or equal to 40 ml/min/1.73m^2 unless lymphoma related
* Prothrombin time/INR (PT) and activated partial thromboplastin time (aPTT) must be < 1.5 x the upper limit of the normal range (ULN); except if, in the opinion of the Investigator, the aPTT is prolonged because of a positive Lupus Anticoagulant.
* Women of childbearing potential must have a negative pregnancy test upon study entry. This is not required for women who are of non-reproductive potential (i.e., post-menopausal by history - defined as: no menses for greater than or equal to 1 year; OR, history of hysterectomy; OR, history of bilateral tubal ligation; OR, history of bilateral oophorectomy).
* The effects of ibrutinib and TEDDI-R on the developing human fetus are unknown. For this reason, women must agree to use highly effective methods of birth control. A "highly effective method of birth control" is defined as a method that has a low failure rate (i.e., less than 1% per year) when used consistently and correctly and includes implants, injectables, birth control pills with two hormones, some intrauterine devices (IUDs). Men who can father children cannot use highly effective methods and are required to use barrier. The specific guidelines are as follows:

  * Women of childbearing potential (WOCBP) must use a highly effective method of birth control and a barrier method, or sexual abstinence (which is defined as refraining from all aspects of sexual activity), while taking the study treatment, as well as for 12 months after the last dose of rituximab.
  * Men who can father children must use a barrier method to prevent pregnancy of their partner and should also not donate sperm while taking the study treatment and for 12 months after the last dose of rituximab.
* Ability of participant or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Systemic chemotherapy less than or equal to 14 days prior to ibrutinib window study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib or other agents used in study
* Participants who are allergic to isavuconazole or any of its ingredients
* Participants who received a strong cytochrome P450 (CYP) 3A inhibitor or inducer within 7 days prior to the first dose of protocol anti-fungal prophylaxis, or participants who require continuous treatment with a strong CYP3A inhibitor/inducer (i.e., with the exception of any medication to be specifically studied in this protocol).

NOTE: In addition, because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list; medical reference texts such as the Physicians Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.

* HIV positive participants will be excluded because of their increased susceptibility to fungal infections which outweighs the potential benefit of participation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or an infection requiring systemic antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Recent infections requiring systemic treatment need to have completed therapy >14 days before the first dose of study drug.
* Pregnant and nursing women are excluded from this study. Pregnant women are excluded in this study because ibrutinib is a tyrosine kinase inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ibrutinib, nursing should be discontinued if the mother is treated with ibrutinib.
* Presence of transfusion-dependent thrombocytopenia.
* History of prior malignancy, with the exception of the following:

  * Malignancy treated with curative intent and with no evidence of active disease present for more than 2 years prior to screening and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanomatous skin cancer or lentigo malignant melanoma without current evidence of disease
  * Adequately treated carcinoma in situ without current evidence of disease.
* Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification, or history of myocardial infarction unstable angina, or acute coronary syndrome within 6 months prior to enrollment in the study.
* Unable to swallow capsules, or disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, or symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* Serologic status reflecting active hepatitis B or C infection. Participants that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. Those who are (PCR positive will be excluded.) Those with a negative PCR for hepatitis B will be treated with antivirals designed to prevent hepatitis B reactivation (e.g., entecavir) and have monitoring for hepatitis B reactivation with PCR.
* History of stroke or intracranial hemorrhage within 3 months prior to enrollment.
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the Investigator s opinion, could compromise the participant s safety, or put the study at undue risk. Participants with suspicious radiologic evidence of aspergillosis infection (i.e., Chest CT and/or Brain MRI) will not be eligible unless confirmatory laboratory testing of Beta-D glucan and aspergillus antigen are negative.
* Concomitant use of warfarin or other vitamin K antagonists within the last 7 days.
* Concurrent systemic immunosuppressant therapy other than corticosteroids (e.g., cyclosporine A, tacrolimus, etc.) within 28 days of the first dose of study drug.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to grade less than or equal to1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia.
* Known bleeding disorders (e.g., von Willebrand s disease) or hemophilia.
* Unwilling or unable to participate in all required study evaluations and procedures.
* Currently active, clinically significant hepatic impairment (greater than or equal to moderate hepatic impairment according to the NCI/Child Pugh classification

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | every 3-6 months
  time from study enrollment until disease progression or death from any cause by arm

SECONDARY OUTCOMES:
Safety and tolerability of TEDDI-R and TEDD-R in sCNSL | ongoing
  the proportion of patients with adverse events leading to discontinuation of therapy
Best overall response after 14 days of ibrutinib monotherapy in sCNSL; after up to 4 cycles of TEDDI-R; and, after up to 4 cycles of TEDD-R (no ibrutinib) | after 14 days and 4 cycles
  proportion of patients who achieve at least a partial response (PR) to therapy
Duration of response (DOR) | every 2 cycles during treatment; every 3-6 months in follow-up
  time from first documentation of tumor response to disease progression
Assessment of pharmacokinetics (PK) and safety of TEDDI-R with concomitant anti-fungal prophylaxis | at least each cycle, up to cycle 4
  time from study enrollment until disease progression or death from any cause
Overall survival (OS) to TEDDI-R and TEDD-R in sCNSL | every 3-6 months
  time from study enrollment until death from any cause
Overall analysis of PFS by arm | every 2 cycles during treatment; every 3-6 months in follow-up
  time from first documentation of tumor response to disease progression
Safety and tolerability of TEDDI-R and TEDD-R in sCNSL by Arm | ongoing
  the proportion of patients with adverse events leading to discontinuation of therapy between arms

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Lakhotia, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@In addition all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. @@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0103.html